CLINICAL TRIAL: NCT02641587
Title: A Randomized, Controlled, Open-label, 2-arm Parallel Group, Single Center Study to Demonstrate Reductions in Exposure to Selected Smoke Constituents in Healthy Smokers Switching to the Carbon Heated Tobacco Product 1.2 (CHTP 1.2), Compared to Continuing to Use Combustible Cigarettes, for 5 Days in Confinement Followed by 85 Days in an Ambulatory Setting.
Brief Title: Reduced Exposure Study Using the CHTP 1.2 With 5 Days in a Confinement Setting Followed by 85 Days in an Ambulatory Setting.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P2R-REXA-07-EU
Record Dates: First submitted 2015-12-23; First posted 2015-12-29 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Smoking
Keywords: Smoking; Cigarettes; Reduced exposure; Confinement; Ambulatory; Carbon Heated Tobacco Product
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHTP 1.2 (Experimental): Ad libitum use of the CHTP 1.2
  Interventions: Other: CHTP 1.2
- CC (Active Comparator): Ad libitum use of subject's own preferred non-menthol brand of CC
  Interventions: Other: CC

INTERVENTIONS:
Other: CHTP 1.2 — Ad libitum use of the CHTP 1.2 for 5 days in confinement followed by 85 days in an ambulatory setting.
  Arms: CHTP 1.2
Other: CC — Ad libitum use of subject's own preferred non-menthol brand of CC for 5 days in confinement followed by 85 days in an ambulatory setting.
  Arms: CC

SUMMARY:
The overall goal of the study is to demonstrate reduction in the levels of biomarkers of exposure (BoExp) to selected harmful and potentially harmful constituents (HPHCs) identified in cigarettes and to obtain safety information in healthy adult smokers switching to the Carbon Heated Tobacco Product 1.2 (CHTP 1.2) as compared to subjects continuing smoking cigarettes (CC) in a confinement setting for 5 days (exclusive use) followed by an ambulatory setting of 85 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged ≥ 28 years.
* Subject is Caucasian.
* Subject is healthy, as judged by the Investigator.
* Subject has smoked at least 10 commercially available non-menthol CCs per day (no brand restrictions) at least for the last 6 weeks prior to the screening visit and admission.
* Subject has smoked at least for the last 10 years.
* Subject does not plan to quit smoking in the next 6 months.

Exclusion Criteria:

* As per Investigator judgment, the subject cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason).
* Subject has received medication within 14 days or within 5 half-lives of the medication (whichever is longer), which has an impact on cytochrome P450 1A2 (CYP1A2) or cytochrome P450 2A6 (CYP2A6) activity.
* Female subject is pregnant or breast feeding.
* Female subject does not agree to use an acceptable method of effective contraception.

Min Age: 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.; Monika Tomaszewska-Kiecana, MD, Principal Investigator — BioVirtus Research Site
Locations (1):
- BioVirtus Research Site Sp. z o.o., Nadarzyn, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bosilkovska M, Tran CT, de La Bourdonnaye G, Taranu B, Benzimra M, Haziza C. Exposure to harmful and potentially harmful constituents decreased in smokers switching to Carbon-Heated Tobacco Product. Toxicol Lett. 2020 Sep 15;330:30-40. doi: 10.1016/j.toxlet.2020.04.013. Epub 2020 May 5. PMID 32380119

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following enrollment of 121 subjects, each subject received a product test of CHTP 1.2 prior to randomization.
  One subject was not randomized due to the physician's decision. This subject is included in the "Exposed Not Randomized" reporting group of the Baseline Characteristics.
  Consequently, 120 subjects were randomized.
Groups:
- Cigarettes (CC): Ad libitum use of subject's own preferred non-menthol brand of CC
  CC: Ad libitum use of subject's own preferred non-menthol brand of CC for 5 days in confinement followed by 85 days in an ambulatory setting.
Period: Confinement Period
Arm/Group | CHTP 1.2 | Cigarettes (CC)
Started | 80 | 40
Completed | 77 | 39
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Period: Ambulatory Period
Arm/Group | CHTP 1.2 | Cigarettes (CC)
Started | 77 | 39
Completed | 76 | 39
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Overall safety population refers to all subjects who were exposed and randomized or exposed and not randomized.
Groups:
- Exposed Not Randomized: "Exposed not randomized" refers to all subjects exposed to CHTP 1.2 but not randomized.
- Total: Total of all reporting groups
Arm/Group | CHTP 1.2 | Cigarettes (CC) | Exposed Not Randomized | Total
Number analyzed (Participants) | 80 | 40 | 1 | 121
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.9 (8.9) | 39.0 (8.0) | 28 | 38.8 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 20 | 1 | 57
  Male | 44 | 20 | 0 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 80 | 40 | 0 | 120
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m2] | 25.74 (3.51) | 25.70 (2.96) | 21.7 | 25.69 (3.33)

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of Monohydroxybutenylmercapturic Acid (MHBMA)
Description: Concentrations measured at Day 5 in urine, adjusted for creatinine.
  Geometric least squares (LS) means and confidence intervals (Cls) from a generalized linear model conducted on log-transformed Day 5 values with log-transformed baseline value, study arm, sex and CC consumption reported at admission as fixed effect factors.
Time Frame: 5 days
Population: Per Protocol (PP) population
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | CHTP 1.2 | Cigarettes (CC)
Number analyzed (Participants) | 74 | 34
pg/mg creat | 285.5 [258.0 to 315.8] | 1904 [1641 to 2209]
Statistical Analysis 1: Comparison: CHTP 1.2 vs Cigarettes (CC); Analysis will be conducted on the natural log scale. The Day 5 levels of MHBMA will be analyzed by means of a generalized linear model using randomized arm as covariate adjusting for sex, average cigarette consumption over the previous 6 weeks prior to Admission (value at Admission for stratification), and log-transformed baseline value of MHBMA; Test type: Other — The analysis will test if the geometric LS mean level of MHBMA for CHTP is lower than for CC. The following hypothesis will be evaluated: H0: XCHTP - XCC ≤ 0.0 HA: XCHTP - XCC > 0.0 where XCHTP and XCC are the geometric LS means of CHTP and CC, respectively. H0 is rejected with a type I error α = 2.5% (one-sided test); p < 0.001, Generalized linear model — The primary endpoints will be tested using a multiple testing procedure to preserve the overall alpha level by simultaneously testing the endpoints using a closed procedure with each test performed at an alpha level of 2.5% one sided; LS Mean Reduction = 85.01, 95% CI 2-sided [82.06 to 87.47] — Least squares (LS) means and estimate of the difference, and 95% CI will be back-transformed for obtaining geometric LS means for each arm, the reduction (calculated as 100% - ratio of CHTP 1.2 : CC [%]), and their 95% CI

2. Primary Outcome: Concentration of 3-hydroxypropylmercapturic Acid (3-HPMA)
Description: as for outcome 1
Time Frame: 5 days
Population: Per Protocol (PP) population
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/mg creat
Arm/Group | CHTP 1.2 | Cigarettes (CC)
Number analyzed (Participants) | 74 | 34
ng/mg creat | 616.8 [565.6 to 672.8] | 1031 [907.9 to 1172]
Statistical Analysis 1: Comparison: CHTP 1.2 vs Cigarettes (CC); Analysis will be conducted on the natural log scale. The Day 5 levels of 3-HPMA will be analyzed by means of a generalized linear model using randomized arm as covariate adjusting for sex, average cigarette consumption over the previous 6 weeks prior to Admission (value at Admission for stratification), and log-transformed baseline value of 3-HPMA; Test type: Other — The analysis will test if the geometric LS mean level of 3-HPMA for CHTP is lower than for CC. The following hypothesis will be evaluated: H0: XCHTP - XCC ≤ 0.0 HA: XCHTP - XCC > 0.0 where XCHTP and XCC are the geometric LS means of CHTP and CC, respectively. H0 is rejected with a type I error α = 2.5% (one-sided test); p < 0.001, Generalized linear model — [p-value comment as in outcome 1, analysis 1]; LS Mean Reduction = 40.20, 95% CI 2-sided [30.25 to 48.73] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Concentration of S-phenylmercapturic Acid (S-PMA)
Description: as for outcome 1
Time Frame: 5 days
Population: Per Protocol (PP) population
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | CHTP 1.2 | Cigarettes (CC)
Number analyzed (Participants) | 74 | 34
pg/mg creat | 386.6 [358.7 to 416.7] | 2401 [2151 to 2681]
Statistical Analysis 1: Comparison: CHTP 1.2 vs Cigarettes (CC); Analysis will be conducted on the natural log scale. The Day 5 levels of S-PMA will be analyzed by means of a generalized linear model using randomized arm as covariate adjusting for sex, average cigarette consumption over the previous 6 weeks prior to Admission (value at Admission for stratification), and log-transformed baseline value of S-PMA; Test type: Other — The analysis will test if the geometric LS mean level of S-PMA for CHTP is lower than for CC. The following hypothesis will be evaluated: H0: XCHTP - XCC ≤ 0.0 HA: XCHTP - XCC > 0.0 where XCHTP and XCC are the geometric LS means of CHTP and CC, respectively. H0 is rejected with a type I error α = 2.5% (one-sided test); p < 0.001, Generalized linear model — [p-value comment as in outcome 1, analysis 1]; LS Mean Reduction = 83.90, 95% CI 2-sided [81.61 to 85.90] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Levels of Carboxyhemoglobin (COHb)
Description: % COHb blood measurements performed in the evening of Day 5, expressed as % of saturation of hemoglobin.
  Geometric least squares (LS) means and confidence intervals (Cls) from a generalized linear model conducted on log-transformed Day 5 values with log-transformed baseline value, study arm, sex and CC consumption reported at admission as fixed effect factors.
Time Frame: 5 days
Population: Per Protocol (PP) population
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: % of saturation of hemoglobin
Arm/Group | CHTP 1.2 | Cigarettes (CC)
Number analyzed (Participants) | 58 | 22
% of saturation of hemoglobin | 2.01 [1.86 to 2.16] | 4.53 [4.01 to 5.11]
Statistical Analysis 1: Comparison: CHTP 1.2 vs Cigarettes (CC); Analysis will be conducted on the natural log scale. The Day 5 levels of COHb will be analyzed by means of a generalized linear model using randomized arm as covariate adjusting for sex, average cigarette consumption over the previous 6 weeks prior to Admission (value at Admission for stratification), and log-transformed baseline value of COHb; Test type: Other — The analysis will test if the geometric LS mean level of COHb for CHTP is lower than for CC. The following hypothesis will be evaluated: H0: XCHTP - XCC ≤ 0.0 HA: XCHTP - XCC > 0.0 where XCHTP and XCC are the geometric LS means of CHTP and CC, respectively. H0 is rejected with a type I error α = 2.5% (one-sided test); p < 0.001, Generalized linear model — [p-value comment as in outcome 1, analysis 1]; LS Mean Reduction = 55.74, 95% CI 2-sided [49.03 to 61.56] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Concentrations of Total 4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol (Total NNAL)
Description: Concentrations measured at Day 90 in urine, adjusted for creatinine.
  Geometric least squares (LS) means and confidence intervals (Cls) from a generalized linear model conducted on log-transformed Day 90 values with log-transformed baseline value, study arm, sex and CC consumption reported at admission as fixed effect factors.
Time Frame: 90 days
Population: Per Protocol (PP) population
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | CHTP 1.2 | Cigarettes (CC)
Number analyzed (Participants) | 57 | 35
pg/mg creat | 37.26 [31.39 to 44.24] | 180.6 [144.8 to 225.1]
Statistical Analysis 1: Comparison: CHTP 1.2 vs Cigarettes (CC); Analysis will be conducted on the natural log scale. The Day 5 levels of Total NNAL will be analyzed by means of a generalized linear model using randomized arm as covariate adjusting for sex, average cigarette consumption over the previous 6 weeks prior to Admission (value at Admission for stratification), and log-transformed baseline value of Total NNAL; Test type: Other — The analysis will test if the geometric LS mean level of Total NNAL for CHTP is lower than for CC. The following hypothesis will be evaluated: H0: XCHTP - XCC ≤ 0.0 HA: XCHTP - XCC > 0.0 where XCHTP and XCC are the geometric LS means of CHTP and CC, respectively. H0 is rejected with a type I error α = 2.5% (one-sided test); p < 0.001, Generalized linear model — [p-value comment as in outcome 1, analysis 1]; LS Mean Reduction = 79.36, 95% CI 2-sided [72.73 to 84.39] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signature of the Informed Consent Form (ICF) until the end of the safety follow-up period, which covered a period of between 128 to 169 days for each subject.
Groups:
- Product Test: After all inclusion/exclusion criteria were checked, all eligible subjects were enrolled and performed a product test using up to five CHTP 1.2
- CHTP 1.2 Confinement: Ad libitum use of the CHTP 1.2 for 5 days in confinement.
- CC Confinement: Ad libitum use of subject's own preferred non-menthol brand of CC for 5 days in confinement.
- CHTP 1.2 Ambulatory: Ad libitum use of the CHTP 1.2 for 85 days in an ambulatory setting.
- CC Ambulatory: Ad libitum use of subject's own preferred non-menthol brand of CC for 85 days in an ambulatory setting.
- CHTP 1.2 Safety FU: CHTP 1.2 Safety Follow-Up period of 28 days
- CC Safety FU: CC Safety Follow-Up period of 28 days
- CHTP 1.2 Post-Randomization: CHTP 1.2 Post-Randomization period
- CC Post-Randomization: CC Post-Randomization period
Arm/Group | Product Test | CHTP 1.2 Confinement | CC Confinement | CHTP 1.2 Ambulatory | CC Ambulatory | CHTP 1.2 Safety FU | CC Safety FU | CHTP 1.2 Post-Randomization | CC Post-Randomization
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/80 | 0/40 | 0/77 | 0/39 | 0/80 | 0/40 | 0/80 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/121 | 1/80 | 0/40 | 1/77 | 1/39 | 0/80 | 0/40 | 2/80 | 1/40
Other Adverse Events (participants affected / at risk) | 62/121 | 37/80 | 12/40 | 50/77 | 26/39 | 1/80 | 1/40 | 64/80 | 31/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Product Test (N=121) | CHTP 1.2 Confinement (N=80) | CC Confinement (N=40) | CHTP 1.2 Ambulatory (N=77) | CC Ambulatory (N=39) | CHTP 1.2 Safety FU (N=80) | CC Safety FU (N=40) | CHTP 1.2 Post-Randomization (N=80) | CC Post-Randomization (N=40)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonsillar Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint Dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Product Test (N=121) | CHTP 1.2 Confinement (N=80) | CC Confinement (N=40) | CHTP 1.2 Ambulatory (N=77) | CC Ambulatory (N=39) | CHTP 1.2 Safety FU (N=80) | CC Safety FU (N=40) | CHTP 1.2 Post-Randomization (N=80) | CC Post-Randomization (N=40)
Headache (Nervous system disorders) | 42 (54) | 9 (10) | 4 (7) | 14 (15) | 8 (9) | 0 (0) | 0 (0) | 20 (25) | 11 (16)
Nasopharyngitis (Infections and infestations) | 3 (3) | 6 (6) | 2 (2) | 9 (9) | 1 (1) | 0 (0) | 0 (0) | 14 (15) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 0 (0) | 14 (15) | 4 (4) | 0 (0) | 0 (0) | 15 (17) | 4 (4)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 8 (8) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 5 (5) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 6 (6) | 3 (3)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 1 (1)
Blood Triglycerides Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
(Gastrointestinal disorders) | 2 (2) | 9 (9) | 2 (2) | 6 (6) | 2 (2) | 0 (0) | 1 (3) | 12 (15) | 5 (7)
Vessel Puncture Site Bruise (General disorders) | 6 (6) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
(Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
(Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
General disorders (General disorders) | 6 (6) | 6 (6) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 7 (7) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specify that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belong to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2016-12-05): https://cdn.clinicaltrials.gov/large-docs/87/NCT02641587/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT02641587/SAP_001.pdf